CLINICAL TRIAL: NCT02189928
Title: Lower Limb Ischaemic Per-conditioning in Acute Cerebral Infarction (<H6): Multicenter Randomized Study With Stratification on IV Thrombolysis and PROBE Design (Prospective Randomized Open Trial With Blinded End-Point)
Brief Title: REmote iSchemic Conditioning in acUtE BRAin INfarction Study
Acronym: RESCUE-BRAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Versailles Hospital (Other)
Collaborators: Unité de Recherche Clinique Paris IDF Ouest (Unknown)
Responsible Party: Principal Investigator, Pr Fernando PICO, Investigator coordinator, Versailles Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P14/01_RESCUE BRAIN; 2014-A00104-43 (Registry Identifier: ID RCB)
Record Dates: First submitted 2014-06-10; First posted 2014-07-15 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Cerebral Infarction
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With per-CID protocol (Experimental): Usual care patients (thrombolysis or not ) with remote ischemic per-conditioning using an electronic tourniquet .
  Interventions: Device: Lower limb tourniquet
- Without per-CID protocol (Other): Usual care patients (thrombolysis or not).
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Lower limb tourniquet — Lower limb tourniquet will be put on half thigh. The protocol will include 4 cycles of inflation cuff 110 mm Hg above systolic blood pressure followed by 4 cycles of deflation in between.
  The total duration of per-CID protocol will be 40 minutes (4 phases of 5 minutes inflations' of and 4 phases of 5 minutes deflations').
  Arms: With per-CID protocol
Other: Usual care
  Arms: Without per-CID protocol

SUMMARY:
Cerebral infarction is the most common form of stroke (80% of strokes). Stroke is the first cause of acquired disability, and the 2nd cause of dementia and death. The only approved treatment in the first 4.5 hour is intravenous rt-PA thrombolysis (Actilyse ®) whose objective is recanalization of occluded artery and reperfusion of the brain parenchyma. Few patients are treated (1-5%) and they keep disability in 50-60% of cases. This handicap is mainly correlated to the final infarct size. The objective of neuroprotective treatments is to reduce the final size of the cerebral infarction.

The per-conditioning remote ischemic (Per-CID) showed a neuroprotective effect in cerebral ischemia by reducing the final size of cerebral infarction animal models. The per-CID corresponds, in cases of cerebral ischemia, to iterative ischemia realization of a member with a cuff. In humans, the per-CID has shown a cardioprotective effect in a randomized control trial involving 250 patients within 6 first hours of myocardial infarction and candidate for primary angioplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Carotid ischemic stroke
* NIHSS score between 5 and 25
* Brain MRI performed within 6 hours from symptoms onset
* Obtaining a written informed consent of the patient or a third party (parent or close), or emergency inclusion process
* Affiliated with a Medicare (or rightful beneficiary)

Exclusion Criteria:

* Presence of a leg ulcer or a bad skin condition in the lower limbs
* History of arterial occlusive disease of the lower limbs
* Sickle cell disease known (risk of vaso-occlusive crisis)
* History of phlebitis in the lower limbs
* History of cerebral infarction older than 3 months
* Participation in another interventional acute phase protocol
* Patients under guardianship
* Pathologies involving life-threatening within 6 months and making it impossible to evaluate to 3 months
* Patient non-self before the ischemic stroke (Rankin Score previous> 2)
* Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Brain MRI changes of DWI ( Diffusion-Weighted Imaging) brain infarction volume (cc) between baseline (<H6) and day 1 in the 2 groups of patients ( Remote Ischemic Perconditioning and control) | 24 hours
  Central lecture of brain MRI, blinded to clinical data, randomisation group and day of MRI realization ( day 0 or day 1) Endpoint criteria: DWI volume d1-d0 (cc) measured by a dedicated software (Neurinfarct) Comparison of DWI volume d1-d0 between the 2 groups ( Per-CID group and control)

SECONDARY OUTCOMES:
Percentage of patients with Modified Rankin Scale (mRS) <2 at 3 months in the 2 groups (PerCID and control) | 3 months
  Percentage of patients with Modified Rankin Scale (mRS) <2 ( i.e. favorable outcome with no disability) at 3 months in the 2 groups (PerCID and control)

OTHER OUTCOMES:
safety of remote perconditioning ischemic process | 7 days
  - Rate of lower limb ischemia and deep venous thrombosis in Per CID group
safety of remote perconditioning ischemic process | 7 days
  Rate of early neurological worsening (NIHSS score (d1- d0) > 4 points) in Per-CID and control group
safety of remote perconditioning ischemic process | 7 days
  Percentage of hemorrhagic transformation in case of IV thrombolysis in the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Fernando PICO, Neurology Department head, Principal Investigator — Versailles Hospital
Locations (9):
- France (9):
  - Centre Hospitalier Sud Francilien, Corbeil-Essonne
  - Hôpital Henri Mondor, Créteil
  - Centre Hospitalier de Versailles, Le Chesnay
  - CHU de Nantes, Nantes
  - Hôpital Pitie-Salpêtrière, Paris
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - Hôpital Bichat, Paris
  - CHU de Strasbourg, Strasbourg
  - Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pico F, Lapergue B, Ferrigno M, Rosso C, Meseguer E, Chadenat ML, Bourdain F, Obadia M, Hirel C, Duong DL, Deltour S, Aegerter P, Labreuche J, Cattenoy A, Smadja D, Hosseini H, Guillon B, Wolff V, Samson Y, Cordonnier C, Amarenco P. Effect of In-Hospital Remote Ischemic Perconditioning on Brain Infarction Growth and Clinical Outcomes in Patients With Acute Ischemic Stroke: The RESCUE BRAIN Randomized Clinical Trial. JAMA Neurol. 2020 Jun 1;77(6):725-734. doi: 10.1001/jamaneurol.2020.0326. PMID 32227157
- [Derived] Pico F, Rosso C, Meseguer E, Chadenat ML, Cattenoy A, Aegerter P, Deltour S, Yeung J, Hosseini H, Lambert Y, Smadja D, Samson Y, Amarenco P. A multicenter, randomized trial on neuroprotection with remote ischemic per-conditioning during acute ischemic stroke: the REmote iSchemic Conditioning in acUtE BRAin INfarction study protocol. Int J Stroke. 2016 Oct;11(8):938-943. doi: 10.1177/1747493016660098. Epub 2016 Jul 19. PMID 27412192